CLINICAL TRIAL: NCT02937948
Title: Phase II Study of Adaptative Radiotherapy for Locally Advanced Cervical Cancer
Brief Title: Adaptative Radiotherapy for Locally Advanced Cervical Cancer
Acronym: ARCOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-02-45-01
Record Dates: First submitted 2016-10-13; First posted 2016-10-19 (Estimated); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Uterine Cervical Cancer
Keywords: Locally advanced
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adaptative Treatment plans (Experimental): A Library of treatment plans will be generated for each patient before starting radiochemotherapy (standard treatment). This Library will be created using CT-Scans with variable bladder filling (and hence different uterine positions). Each day of radiotherapy treatment, an appropriate plan is chosen based on Imaging that day.
  Interventions: Other: Adaptative treatment plan; Radiation: External radiotherapy

INTERVENTIONS:
Other: Adaptative treatment plan — Each patient will have 3 scanners before treatment initiation. One corresponding to an empty bladder, one to an "intermediate" one, one to a full bladder.
Radiation: External radiotherapy — At the time of each fraction of external radiotherapy, the most appropriate plan (empty, intermediate, full bladder) covering the target and sparing the organs at risk is chosen.

SUMMARY:
This study evaluates the effect of adaptative Intensity-Modulated Radiation Therapy (IMRT) in the treatment of locally advanced cervical cancer on acute genito-urinary (GU), and gastrointestinal (GI) toxicities. Every patients will be treated according to the adaptative IMRT strategy.

ELIGIBILITY:
Inclusion Criteria:

* Cervix carcinoma proved by histology
* According International Federation of Gynecology and Obstetrics (FIGO) classification, stages IB2, IIA, IIB, IIIA and IIIB without lumbo-aortic lymph node damage (surgical or radiologic)
* Patient treated with radio-chemotherapy then curietherapy with curative aim, validated in multidisciplinary meeting
* Renal, hepatic and cardiovascular functions that allow administration of the associated systemic treatment
* Older than 18 years
* Good general status, World Health Organization less or equal to 1
* Signed informed consent

Exclusion Criteria:

* History of cancer that is not controlled and / or treated for less than 5 years (excepted for cutaneous baso-cellular cancer)
* History of pelvic irradiation
* Simultaneous participation to another research that could interfere with the study results
* Pregnant or breastfeeding patient
* Patient under tutor or guardian
* Patient not able to respect medical follow-up for geographical, social or psychological reasons
* Not affiliated to a system of French social security

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Number of patient having an Acute genito-urinary (GU) and Gastro-intestinal (GI) toxicities assessed by CTCAE V4.03 | 3 months after end of radio-chemotherapy treatment

SECONDARY OUTCOMES:
Number of patient having a Grade ≥ 2 Hematologic and other toxicities assessed by CTCAE V4.03 | 3 months after end of radio-chemotherapy treatment

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - Institut de Cancérologie de l'Ouest, Angers
  - Centre François Baclesse, Caen
  - CLCC Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Centre rené Gauducheau, Nantes
  - CHU Poitiers, Poitiers
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - CHU de Tours, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
Not authorized in France